CLINICAL TRIAL: NCT00330200
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Examine the Effects of ISIS 113715 Monotherapy on Insulin Sensitivity, Glucose and Lipid Metabolism and Energy Expenditure in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effects of ISIS 113715 on Insulin Sensitivity, Glucose, and Lipid Metabolism and Energy Expenditure in Type 2 Diabetics
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor enrollment
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Isis Pharmaceuticals, Isis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 113715-CS11
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2008-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Fasting plasma glucose; HbA1c; Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ISIS-113715

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ISIS 113715

SUMMARY:
The aim of this study is to examine the effects of ISIS 113715 monotherapy on insulin sensitivity, glucose and lipid metabolism and energy expenditure in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (post menopausal and/or surgically sterile)
* Aged 18 to 70 years
* Treatment naïve subjects with fasting blood glucose levels of 150-220 mg/dL, hematocrit of >/= 35% and HbA1c levels of >/= 7% and </= 10.0%
* Subjects on antidiabetic therapy with fasting blood glucose levels of 100-200 mg/dL, hematocrit of >/= 35%, and HbA1c levels of >/= 6.5% and </= 9.0%

Exclusion Criteria:

* Greater than 3 severe hypoglycemic episodes within six months of screen
* Pregnant, breastfeeding, or intends to become pregnant
* Clinical signs or symptoms of liver disease, acute or chronic hepatitis, or ALT greater than 1.5 times the upper limit of normal
* History of hepatitis B surface antigen, hepatitis C antibody, or HIV
* Complications of diabetes (e.g., neuropathy, nephropathy, and retinopathy)
* Clinically significant and currently active diseases
* Clinically significant abnormalities in medical history, physical examination, or laboratory examination

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2007-03-01 (Actual); Study Completion 2007-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of ISIS 113715 on hepatic and peripheral insulin sensitivity
Examine the effect on whole body energy expenditure
Evaluate the effects on fasting and postprandial glucose excursions
Evaluate the effects on hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Expand the safety and tolerability profile for ISIS 113715
Assess the effects of ISIS 113715 on rates of basal and insulin stimulated whole body glycerol turnover
Assess the effects of ISIS 113715 on insulin suppression of local rates of lipolysis (microdialysis)

CONTACTS AND LOCATIONS:
Overall Officials: Isis Pharmaceuticals, Study Chair — Ionis Pharmaceuticals, Inc.
Locations (1):
- Yale - New Haven Hospital, New Haven, Connecticut, United States